CLINICAL TRIAL: NCT04977466
Title: NIH Intramural Research Program's Pregnancy Registry Protocol for Subjects and Their Partners
Brief Title: NIH Intramural Research Program s Pregnancy Registry Protocol for Subjects and Their Partners
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10000268; 000268-CC
Record Dates: First submitted 2021-07-24; First posted 2021-07-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Pregnancy Outcome
Keywords: Partner; Intramural Research Program; OFFSPRING; Registry; Delivery; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group #1 / Pregnant Female NIH Participants: Female NIH study participants.
- Group #2 / Male and Female Partners: Male or female partners of women who participated in NIH intramural clinical trials and that became pregnant.
- Group #3 / Pregnant Female Partners of Male or Female NIH Clinical Trial Partici: Female partners of NIH intramural clinical trial participants who became pregnant while their partner was or within 1 year after the last day of intervention after their partner was on a study.
- Group #4 / Neonate or Offspring of a Pregnant Female Participant or Pregnant Fe: Offspring from birth to 12 months of age and born to female participants / female partners.

SUMMARY:
Background:

In 2018, the NIH intramural research program had almost 23,000 people taking part in active clinical research studies. Half of those people were female. More than a third were of child-bearing age. Researchers want to use data from this group to create a pregnancy registry. It will be used to collect data about pregnancy and birth outcomes related to unplanned exposure to research products. These products may include drugs, vaccines, treatments, and interventions.

Objective:

To collect data about pregnancies and births from people who took part in an NIH clinical trial and their partners who became pregnant while in the study or shortly after.

Eligibility:

People of any age and their partners who took part in an NIH clinical trial and became pregnant while in the study or within 1 year after.

Design:

Participants will be screened by phone. Their clinical trial history will be verified.

Participants will be interviewed in person, by phone, or virtually. They will be asked about their health and their trial experience in relation to their pregnancy. They will give details about their pregnancy and baby (if appliable). They will be interviewed every 6 months for 1 year after the birth of their baby, as applicable.

Data from both NIH and outside medical records will be used. Participants will give their doctor s name and contact details. They will provide a release for their records to be used. If needed, they will provide a release for their baby s records.

Data will be coded and stored in a database on an in-house NIH secure server. Data may be used in future studies

DETAILED DESCRIPTION:
Study Description:

This protocol will serve as a pregnancy registry to collect prospective and retrospective health information from current and former NIH intramural research participants, their partners and offspring that became pregnant during or within 1 year after participating in an NIH intramural clinical trials. The registry will provide supplemental data on outcomes of clinical trial interventions on pregnancy and delivery of offspring as this information is seldom available because pregnant women are often immediately excluded from study participation upon becoming pregnant and data from women who became pregnant and their offspring outcomes is not systematically or routinely collected and evaluated in the intramural program at the NIH. Partners of women who became pregnant within 1 year following research study participation in clinical trials will be invited to participate to evaluate if participation in clinical trials extends to those in close contact.

Objective:

To collect information about pregnancy and offspring outcomes from NIH intramural clinical trial participants and/or partners of current and former NIH research participants.

Study Population:

Adult participants:

Females that participated in NIH intramural clinical trials and became pregnant while on study or within 1 year after.

Male or female partners of women that participated in NIH intramural clinical trials that became pregnant while they were on study or within 1 year after.

Female partners of NIH intramural clinical trials participants that became pregnant while their partner was or within 1 year after their partner was on a study.

Offspring from birth to 12 months of age and born to:

Females that participated in NIH intramural clinical trials and became pregnant while on study or within 1 year after.

Male or female partners of women that participated in NIH intramural clinical trials that became pregnant while they were on study or within 1 year after.

Female partners of NIH intramural clinical trials participants that became pregnant while their partner was or within 1 year after their partner was on a study.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* All Participants

  * Able and willing to provide written informed consent for study participation.
  * Stated willingness to comply with all data collection study activities
  * Male or female, aged 0-100 years
  * Participant or partner of a participant on NIH protocol
* Group #1 (Pregnant Female NIH Participants)

Female NIH study participants with a confirmed pregnancy that occurred during or within 1 year after the last day of intervention during participation in NIH intramural clinical trials AND that meet at least one of the following criteria/assessments:

* Positive pregnancy test (serum or urine)
* Auscultation of fetal heart tones
* Clinical assessment of fetal movement
* Demonstration of pregnancy by ultrasound

  * Group #2 (Male and Female Partners)

Male or female partners of women who participated in NIH intramural clinical trials and that became pregnant while they were on study or within 1 year of the last day of intervention.

-Group #3 (Pregnant Female Partners of Male or Female NIH Clinical Trial Participants)

Female partners of NIH intramural clinical trial participants who became pregnant while their partner was or within 1 year after the last day of intervention after their partner was on a study AND who meet at least one of the following criteria/assessments:

* Positive pregnancy test (serum or urine)
* Auscultation of fetal heart tones
* Clinical assessment of fetal movement
* Demonstration of pregnancy by ultrasound

  * Group #4 (Neonate or Offspring of a Pregnant Female Participant or Pregnant Female Partner)

Offspring from birth to 12 months of age and born to:

* Females who participated in an NIH intramural clinical trial and became pregnant while on study or within 1 year after.
* Female partners of women or men who participated in an NIH intramural clinical trial who became pregnant while they were on study or within 1 year after.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Participation in NIH research studies that do not meet criteria of a clinical trial, such as natural history or observational studies
* Pregnancy that occurs/occurred more than 1 year after NIH clinical trial participation

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants of NIH IRP protocols.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2045-12-30 (Estimated); Study Completion 2045-12-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment of the last study subject | End of study
  The only outcome of the study is to enroll all study stubjects.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A Guptill, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000268-CC.html